CLINICAL TRIAL: NCT06533085
Title: Comparison Ultrasound-Guided Adductor Canal Block and Surgeon-Performed Block for Pain Management After Total Knee Arthroplasty: A Prospective Randomized Controlled Study
Brief Title: Comparison Ultrasound-Guided Adductor Canal Block and Surgeon-Performed Block for Pain Management After Total Knee Arthroplasty
Acronym: ACB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Fevzi Cakmak, assistant proffesor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-08/89
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthrosis Knee Arthroplasty Analgesia Pain Management
Keywords: Knee Arthroplasty Pain Adductor Canal Block analgesia

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was designed as blinded, randomized and controlled.the person who evaluates the patients before and after the treatment is blind.In other words,the person evaluating the patients and the person giving the treatment are different.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adductor canal block by surgeon (Active Comparator): The method described by Pepper et al. was employed [20]. Accordingly, the anatomical landmarks were first determined by the surgeon post-implantation. The medial femoral cavity was dissected with finger dissection. The vastus medialis obliquus muscle was dissected laterally. The needle was advanced posterior-superiorly by resting it on the anteromedial aspect of the femur at a 45° angle, approximately four finger breadths (7 cm) proximal to the joint line. It was ensured that the needle was not within an artery, and a 22G 10 cm needle was used to inject 7 ml of 0.5% bupivacaine + 8 ml of 0.9% saline. No additional peri-articular injection was performed
  Interventions: Procedure: Adductor canal block by surgeon
- Adductor canal block by anesthesiology specialist (Active Comparator): The anesthesiologist used an ultrasound-guided technique without a stimulator aid to apply the adductor canal block. While the patient was supine, the leg position was done with a slight external thigh rotation.Our target zone for the adductor canal block was the inner mid-thigh, where the vasoadductor membrane can be seen on the medial border of the vastus medialis muscle and the lateral side of the femoral artery. After ultrasonography visualization of the vasoadductor membrane, the needle was targeted to the membranous structure beside the femoral artery. A mixture of 7 ml 0.5% bupivacaine with 8 ml of %0.9 isotonic saline solution was injected slowly into the particular area as peri-articular filling lateral to the femoral artery was seen
  Interventions: Procedure: Adductor canal block by surgeon
- Control group (Active Comparator): The posterior capsular infiltration analgesia procedure was performed following irrigation procedures before implantation. The PCI procedure involves injecting 20 mL of the PCI cocktail (consisting of 0.2% ropivacaine and 2.0 mg/mL epinephrine) into the posterior aspect of the capsule through the intercondylar space of the femur. The PCI cocktail was prepared by an anesthesiologist who was not a part of the study
  Interventions: Procedure: Adductor canal block by surgeon

INTERVENTIONS:
Procedure: Adductor canal block by surgeon — Three groups were evaluated in the study. All three groups underwent intraoperative PCI.
  Group 1 (Adductor canal block by surgeon) Group 2 (Adductor canal block by anesthesiology specialist ) Group 3 (Control group)
  Other Names: Adductor canal block by anesthesiology specialist

SUMMARY:
Objective: Adductor canal block (ACB) is widely performed for postoperative analgesia for total knee arthroplasty (TKA). The aim of this study is to compare surgeon-assisted and anesthesiologist-assisted (ultrasound-guided) adductor blocks in terms of postoperative analgesic efficacy.

Methods: This study was designed as a double-blind, prospective and randomized trial. A total of 240 participants were randomly allocated to three groups: one where the surgeon performed the adductor canal block (ACBs), another where it was conducted by an anesthetist with ultrasound guidance (ACBa), and a third group without the adductor block. The follow-up management after the Total Knee Arthroplasty (TKA) procedure occurred on the first, third, and tenth days, as well as the twelfth week. Outcome measures comprised pain assessment using the Visual Analog Scale (VAS) and monitoring opioid analgesic consumption.

DETAILED DESCRIPTION:
1. Introduction In advanced stages of osteoarthritis (OA) of knee, one of major option of treatment is total knee arthroplasty (TKA). Approximately 20% of individuals who undergo TKA experience a loss of physical function, primarily due to the variable intensity of post-operative pain. The risk of thromboembolism due to ambulation limitations and immobility increases along with pain . Various approaches have been proposed to manage post-operative pain. Three distinct regimens have been developed to control pain that develops after TKA. These can be pre-operative, intraoperative, and post-operative analgesic regimens . The main component of the pre-operative regimen is opioids. Local infiltration analgesic regimens are considered in the intraoperative regime, while peripheral nerve blocks are examined in the post-operative analgesic regime .

   Opioids are effective in pain management, yet they come with limited side effects . Local infiltration anesthesia administration is straightforward and carries a low risk of systemic toxicity . While various methods exist, the posterior capsule is a commonly targeted administration site. Adductor canal block (ACB) can be performed pre-operatively, intraoperatively, or post-operatively. The motor branches of the femoral nerve are preserved while blocking the saphenous nerve, and quadriceps muscle strength is minimally affected. Hospital stay is shortened. ACB is becoming increasingly popular due to these advantages. ACB is routinely performed with ultrasound (USG) pre-operatively or post-operatively. In addition, intraoperative ACB performed by the surgeon has recently been introduced. One of the techniques utilized to alleviate post-operative pain is known as posterior capsular infiltration analgesia (PCI). In PCI, local sensory nerve endings are targeted. PCI preserves muscle strength and does not negatively impact functional recovery.

   The objective of this study is to compare postoperative pain among knee prosthesis patients who undergo adductor canal block (ACBa) performed by an anesthetist using ultrasound guidance, ACB (ACBs) performed intraoperatively by the surgeon, and those without ACB.
2. Materials and Methods This study has been designed in a double-blind, randomized, controlled trial format. The study included 255 participants diagnosed with knee osteoarthritis and underwent TKA surgery between May 2021 and May 2022 at our university hospital. The sample size for the study was determined through a power analysis. Based on power analysis for the F-test with a Type I error rate of 0.05, a 95% confidence interval, and a Type II error rate of 0.10, the requisite total sample size is determined to be 207 subjects (equating to 69 patients per group). Owing to the potential employment of non-parametric tests within the analyses, it is recommended to augment the sample size by 15%. Consequently, the calculated sample size necessary is established at 240 subjects (thereby requiring 80 patients per group). This study will be conducted in accordance with the principles of the Declaration of Helsinki. Ethical approval for the study was been obtained from the ethics committee of the institution where the researchers are employed (Kirsehir Ahi Evran University, Faculty of Medicine Ethics Committee, IRB approval number: 2022-08/89). Participation was voluntary. Informed consent was obtained from the participants, indicating that their information would be used in the study, but their identities would remain confidential.

Physical examinations were repeated on participants before the surgery, and pre-operative anesthesia examinations were conducted. At this stage, the acceptance criteria for the participants were evaluated. Inclusion criteria were defined as end stage (Kellgren-Lawrence grade 4) knee osteoarthritis, treated with primary TKA and willing to participate the study. The following were excluded from the study: refusal to participate, underwent revision TKA, allergy to any of the painkillers used, contraindication to regional or spinal anesthesia, use of narcotic painkillers prior to surgery, sensory or motor neuropathy, cirrhosis of the liver, chronic renal failure. The study was continued with 240 participants after excluding those who did not meet the criteria. The participants were randomly divided into three groups, one being the control group. Figure 1 shows the Consolidated Standards of Reporting Trials (CONSORT) diagram.

A computer-generated randomized list was generated from which participants were randomly allocated to one of the three study groups in a 1:1:1 allocation ratio. Adductor canal block plus posterior capsular infiltration analgesia was performed intra-operatively by the surgeon using anatomical landmarks, and no additional imaging was performed (ACBs). Adductor canal block plus posterior capsular infiltration analgesia was performed post-operatively by a specialist in anesthesiology with the help of ultrasound (ACBa). Finally, a control group underwent PCI only. Patients were evaluated postoperatively by different authors for double-blind.

Participants and the surgeons conducting pre-operative and post-operative assessments need to be made aware of the group to which the patient belongs. The surgeon performing the operation is distinct from the one conducting the assessment.

All participants underwent surgery by a single senior surgeon, under spinal anesthesia performed by a single experienced anesthesiologist. The participants were prepared for the operation by applying lateral support in the supine position under spinal anesthesia. Following the administration of spinal anesthesia, a dose of 10 mg/kg of tranexamic acid was administered intravenously to each patient before the commencement of the surgical procedure. The surgical procedure involved a standard midline skin incision followed by a medial parapatellar arthrotomy. Subsequently, standard tibial and femoral osteotomies were performed with the use of a tourniquet during implant cementation. The Genesis II (Smith & Nephew, Memphis, TN) primary posterior-stabilized implant was utilised. The tourniquet was inflated at the stage when the cuts were completed and the washing procedure began. The implant was then performed, the cement reaction was completed, and the tourniquet cuff was lowered. Total knee arthroplasty with a tourniquet and cement was used in all participants.

Three groups were evaluated in the study. All three groups underwent intraoperative PCI.

Group 1 (Adductor canal block by surgeon): The method described by Pepper et al. was employed. Accordingly, the anatomical landmarks were first determined by the surgeon post-implantation. The medial femoral cavity was dissected with finger dissection. The vastus medialis obliquus muscle was dissected laterally. The needle was advanced posterior-superiorly by resting it on the anteromedial aspect of the femur at a 45° angle, approximately four finger breadths (7 cm) proximal to the joint line. It was ensured that the needle was not within an artery, and a 22G 10 cm needle was used to inject 7 ml of 0.5% bupivacaine + 8 ml of 0.9% saline. No additional peri-articular injection was performed (Figure 2).

Group 2 (Adductor canal block by anesthesiology specialist ): This method was performed post-operatively right after the surgery was over. The anesthesiologist used an ultrasound-guided technique without a stimulator aid to apply the adductor canal block. While the patient was supine, the leg position was done with a slight external thigh rotation. After proper positioning, the skin was prepared with an iodine solution, and a sterile technique was used. For block performance, a 22-gauge 100 mm needle and linear ultrasound probe were chosen. Our target zone for the adductor canal block was the inner mid-thigh, where the vasoadductor membrane can be seen on the medial border of the vastus medialis muscle and the lateral side of the femoral artery. Sartorius muscle was seen anterior to all three of those structures. After ultrasonography visualization of the vasoadductor membrane, the needle was targeted to the membranous structure beside the femoral artery. A mixture of 7 ml 0.5% bupivacaine with 8 ml of %0.9 isotonic saline solution was injected slowly into the particular area as peri-articular filling lateral to the femoral artery was seen (Figure 3).

Group 3 (Control group): The posterior capsular infiltration analgesia procedure was performed following irrigation procedures before implantation. The PCI procedure involves injecting 20 mL of the PCI cocktail (consisting of 0.2% ropivacaine and 2.0 mg/mL epinephrine) into the posterior aspect of the capsule through the intercondylar space of the femur. The PCI cocktail was prepared by an anesthesiologist who was not a part of the study (Figure 4).

Postoperative rehabilitation and management: Continuous physical therapy was conducted to measure the patient's endurance at certain movement degrees. The device was set at 45° on the first day after surgery, and rehabilitation began. Those who tolerated rehabilitation for 60 minutes were gradually increased to 75°, 90°, 105°, and 120°. On the first day, a maximum of 90° was allowed, and on the second day, the 105° and 120° were moved to those who tolerated it. The angle the participants could tolerate and how long was recorded on the 1st, second, and third days. Metamizole sodium 500 mg/dose every 6 hours intravenously, celecoxib (orally, once daily, 400 mg per dose), paracetamol (oral, four times daily, 500 mg per dose), pregabalin (orally, once daily, 75 mg per dose) were given for postoperative pain management. Patient with persisted paint or could not tolerate rehabilitation, single dose (2 ml) containing 100 mg of tramadol hydrochloride was administered.

Examined Variables: The participants' age, gender, body mass index, and the side of the operation were examined. The participants' need and consumption of opioids. (One ampoule (2 ml) contains 100 mg of tramadol hydrochloride. Range of motion (ROM) was measured pre-operatively and 12th week post-operatively. The Knee Society Score (KSS) and the Oxford Knee Score (OKS) were also measured preoperatively and at 12 weeks post-operatively to assess functional status. VAS scores were recorded for the participants before surgery and at 3 h, 12 h, first day, 3 days, 10 days and 12 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Performing total knee joint arthroplasty due to stage 4 gonarthrosis
* Agree to participate in the study
* Having signed the informed consent form

Exclusion Criteria:

* The following were excluded from the study: refusal to participate
* Underwent revision TKA,
* Allergy to any of the painkillers used,
* Contraindication to regional or spinal anesthesia,
* Use of narcotic painkillers prior to surgery,
* Sensory or motor neuropathy,
* Cirrhosis of the liver,
* Chronic renal failure

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | immediately before surgery and postoperative at hour 3, postoperative at hour 12, postoperative day 1, postoperative day 3, postoperative day 10 and week 12 after surgery.
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Managment | Postoperative Day 1 Opioid Usage, Postoperative Day 2 Opioid Usage, Postoperative Day 3 Opioid Usage
  consumption of opioids (single dose (2 ml) containing 100 mg of tramadol hydrochloride was administered)

SECONDARY OUTCOMES:
Functionality | preoperatively and at week 12 post-operatively
  Knee scoiety score(KSS) (The original KSS has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.Turkish validity and reliability has been established.)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahievran university, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cakmak MF, Horoz L, Arslan FN, Demir OU, Basarir K. Comparison ultrasound-guided adductor canal block and surgeon-performed block for pain management after total knee arthroplasty: a prospective randomized controlled study. BMC Musculoskelet Disord. 2024 Aug 10;25(1):637. doi: 10.1186/s12891-024-07762-x. PMID 39127622